CLINICAL TRIAL: NCT02190916
Title: Illness Perception, Fatigue, and Function in Systemic Vasculitis (The VCRC Vasculitis Perception (VIP) Study)
Brief Title: Vasculitis Illness Perception (VIP) Study
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Boston University (Other); Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 5533
Record Dates: First submitted 2014-05-30; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Wegener Granulomatosis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Polyarteritis Nodosa; Giant Cell Arteritis; Takayasu's Arteritis; Henoch-Schoenlein Purpura; Behcet's Disease; CNS Vasculitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Polyarteritis Nodosa; Giant Cell Arteritis; Takayasu Arteritis; IgA Vasculitis; Behcet Syndrome; Vasculitis, Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn about how patients with vasculitis think about their illness and to assess to what extent patient perceptions of illness are associated with physical, mental, and social functioning

DETAILED DESCRIPTION:
All patients enrolled in the Vasculitis Clinical Research Consortium's Contact Registry were invited via email to participate in this study. The Contract Registry includes people who self-identify as having one of the following types of vasculitis: granulomatosis with polyangiitis (Wegener's), microscopic polyangiitis, Churg-Strauss syndrome, polyarteritis nodosa, Takayasu's arteritis, giant cell arteritis, Behcet's disease, Henoch-Schöenlein purpura, or CNS vasculitis. People voluntarily enroll in this Registry with the understanding that they will receive information about clinical studies for which they might be eligible. The introductory email included basic information about the study and all of the required elements for informed consent in a brief format. Once participants agreed to participate in the study, then they were directed to the online questionnaire.

When completing the questionnaire, patients were asked a series of questions. Some of the follow-up questions depended on initial answers. The questionnaire content was included as an appendix. The online questionnaire version was thoroughly tested for usability.

It was expected that most participants would require approximately 20-30 minutes to complete the questionnaire.

The survey data is stored by the Rare Diseases Clinical Research Network Data Management and Coordinating Center (DMCC) at the University of South Florida. The data is de-identified. Names or other personal health information are not be collected.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in VCRC Contact Registry
* Patient reported diagnosis of granulomatosis with polyangiitis (Wegener's granulomatosis), Microscopic Polyangiitis, Churg-Strauss Syndrome, Polyarteritis Nodosa, Giant Cell Arteritis, Takayasu's Arteritis, Henoch-Schöenlein Purpura, Behçets disease, and CNS Vasculitis
* 18 years of age or older
* English speaking

Exclusion Criteria:

* Inability to provide informed consent and complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from within the Vasculitis Clinical Research Consortium (VCRC) Patient Contact Registry to participate in an online questionnaire. More than 2000 patients, representing all the different types of idiopathic vasculitis, are currently enrolled into the on-line registry. The different types of vasculitis available for study include: granulomatosis with polyangiitis (Wegener's granulomatosis), microscopic polyangiitis, Churg-Strauss Syndrome, polyarteritis nodosa, giant cell arteritis, Takayasu's arteritis, Henoch-Schöenlein purpura, Behçets disease, and CNS vasculitis.
Sampling Method: Non-Probability Sample
Enrollment: 707 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Composite measure to include Illness perceptions, fatigue and function in patients with systemic vasculitis with further emphasis on causal beliefs about disease onset and relapse triggers. | 1 year after the study is closed to enrollment
  The outcome measure(s) will be evaluated based on the cross-sectional online questionnaire. The questionnaire is the only study procedure for this online patient contact registry protocol and will be the sole analysis tool for both the primary and secondary outcome measures.

SECONDARY OUTCOMES:
Composite measure of potential associations between illness perceptions, fatigue and function in patients with systemic vasculitis | 1 year after the study is closed to enrollment
  The outcome measure(s) will be evaluated based on the cross-sectional online questionnaire. The questionnaire is the only study procedure for this online patient contact registry protocol and will be the sole analysis tool for both the primary and secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Grayson, MD, Study Chair — Boston University; Lianna Fraenkel, MD, MPH, Study Chair — Yale University; Peter A. Merkel, MD, MPH, Study Chair — Boston University; Naomia A. Amudala, NP, Study Chair — Boston University; Amanda M. Terry, MA, Study Chair — University of South Florida College of Medicine
Locations (1):
- University of South Florida Data Management Coordinating Center, Tampa, Florida, United States